CLINICAL TRIAL: NCT01238497
Title: Edwards SAPIEN™ Aortic Bioprosthesis Multi-Region Outcome Registry XT
Brief Title: SOURCE XT REGISTRY
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-10
Record Dates: First submitted 2010-10-26; First posted 2010-11-10 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Severe Aortic Stenosis
Keywords: SAPIEN XT™; Transfemoral; NovaFlex; NovaFlex+; NF; NF+; Transapical; Transaortic; Ascendra2; Ascendra+; Asc+; aortic stenosis; aortic valve; Transcatheter Heart Valve; THV
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Registry 1 - SOURCE XT: Registry 1: All patients implanted with a SAPIEN XT valve, via Transfemoral access using NovaFlex (for 23mm and 26mm valve), or via Transapical access using Ascendra2 (23mm, 26mm and 29mm valve)
  Interventions: Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis
- Registry 2 - Ascendra+: Registry 2: All patients implanted with a SAPIEN XT Valve, via Transapical or Transaortic access using Ascendra+ delivery system (23mm, 26mm and 29mm valve)
  Interventions: Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis
- Registry 3 - NovaFlex+ 29 mm: Registry 3: All patients implanted with a SAPIEN XT valve, 29mm only, via Transfemoral access using NovaFlex+
  Interventions: Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis

INTERVENTIONS:
Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis — Patients eligible for either transfemoral or transapical access and any of the 3 valve sizes (23, 26 or 29)
  Other Names: TAVI Transcatheter Aortic Valve Implantation
  Groups: Registry 1 - SOURCE XT
Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis — Patients eligible for transapical or transaortic access and any of the 3 valve sizes (23mm, 26mm or 29mm)
  Other Names: TAVI Transcatheter Aortic Valve Implantation
  Groups: Registry 2 - Ascendra+
Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis — Patients eligible for transfemoral access and requiring a 29mm valve.
  Other Names: TAVI Transcatheter Aortic Valve Implantation
  Groups: Registry 3 - NovaFlex+ 29 mm

SUMMARY:
This registry is to expand upon existing data sets, to identify patient characteristics and indicators related to complications and clinical benefits for patients with symptomatic severe calcific degenerative aortic stenosis that are undergoing treatment with the commercially available Edwards SAPIEN XT™ Valve, and delivery devices.

DETAILED DESCRIPTION:
Consecutive patient data should be collected at discharge, 30 days and 12 months post-implant. Subsets of patients may undergo additional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The SAPIEN XT™ THV is indicated for use in patients with symptomatic aortic stenosis requiring TAVI who have a high risk for operative mortality, or are "non-operable"

Exclusion Criteria:

* Non-valvular or congenital aortic stenosis
* Pre-existing prosthetic heart valve in the Aortic position or a non-calcified aortic valve
* Severe (>3+) mitral insufficiency or aortic regurgitation > 3+
* Active bacterial endocarditis or other active infections
* Severe ventricular dysfunction with ejection fraction < 20%
* Coronary artery disease-related unstable angina
* Inability to tolerate anticoagulation / antiplatelet therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 2954 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Assess and track causality and sequelae of major adverse events | 30 days

SECONDARY OUTCOMES:
Effectiveness: observe trends in patient characteristics and outcomes over time | One year

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Wendler, MD, PhD, FRCS, Principal Investigator — olaf.wendler@kch.nhs.uk
Locations (104):
- Austria (2):
  - Universitatsklinik Innsbruck, Innsbruck
  - Medical University Vienna, Vienna
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Clinique St Luc, Bouge
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Services, Hamilton, Ontario
  - Southlake Hospital, Newmarket, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier De Universite of Montreal, Montreal, Quebec
  - Hospital Laval, Sainte-Foy, Quebec
- University of Hradec Kralove, Hradec Králové, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (16):
  - CHU Jean Minjoz, Besançon
  - CHU La Cavalle Blanche, Brest
  - Hôpital Privé Parly II, Le Chesnay
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU La Timone, Marseille
  - Hôpital St Joseph, Marseille
  - Clinique Clairval, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - CHU Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hopital Nord Laënnec, Nantes
  - Hopital Bichat, Paris
  - CHRU Pontchaillou, Rennes
  - C.H.U Charles Nicolle, Rouen
  - CHU Rangueil, Toulouse
  - Clinique Pasteur / GCVI, Toulouse
  - Clinique Saint-Gatien, Tours
- Germany (29):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen GmbH, Bad Krozingen
  - Kerckhoff Klinik, Bad Nauheim
  - Herz- und Gefäss-Klinik GmbH, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, Bad Oyenhausen
  - Evangelisch Freikirchliches Krankenhaus, Bernau
  - Universitätsklinikum, Cologne
  - Städtisches Klinikum, Dortmund
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitätsklinik Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitatsmedizin Gottingen, Göttingen
  - Asklepios Klinik St Georg, Hamburg
  - Universitatsklinikum Eppendorf, Hamburg
  - Universitätsklinikum, Jena
  - KLINIKUM KARLSBURG der Klinikgruppe Dr. Guth GmbH & Co. KG, Karlsburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Herzzentrum Leipzig GmbH, Leipzig
  - Johannes Gutenberg Universität Mainz, Mainz
  - Deutsches Herzzentrum Muenchen, Munich
  - Klinikum Schwabing, Munich
  - Klinikum der Universität München - Großhadern, Munich
  - Klinikum Bogenhausen, Munich
  - Universitätsklinikum Münster, Münster
  - Klinikum Sud Nurnberg, Nuremberg
  - Universitatsklinikum Regensburg, Regensburg
  - SANA Herzzentrum, Stuttgart
  - Universitatsklinik Wurzburg, Würzburg
- Hygeia Hospital, Athens, Greece
- Israel (4):
  - Rambam Medical Center, Haifa
  - Shaare Zedek, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Clinica Sant'Anna Hospital, Catanzaro
  - Ospedale Pasquinucci, Massa
  - Clinica Montevergine, Mercogliano
  - Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino, Milan
  - Hesperia Hospital, Modena
  - Azienda Ospedaliera Policlinico Universitario, Padua
  - Istituto Clinico Humanitas, Rozzano Milano
  - Ospedale San Giovanni Battista, Torino
- Maastricht UMC+, Maastricht, Netherlands
- Universitetssykehuset Nord-Norge, Tromsø, Norway
- The Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw, Poland
- South Africa (5):
  - Sunninghill Hospital, Johannesburg, Gauteng
  - St Augustine's Hospital, Durban
  - Panorama Medi-Clinic, Grand Rapids
  - UNITAS Hospital, Pretoria
  - Vergelegen Medi-Clinic, Somerset West
- Spain (10):
  - C.H.U. A Coruña, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Vall Hebron, Barcelona
  - Policlinica Gipuzkoa, Donostia / San Sebastian
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Virgen de Arrixaca, Murcia
  - Hospital Marques de Valdecilla, Santander
  - Hospital Virgen Macarena, Seville
  - Complexo Hospitalario Universitario de Vigo, Vigo
- Switzerland (2):
  - Inselspital Bern, Bern
  - Klinik im Park, Zurich
- United Kingdom (5):
  - London Chest Hospital, London
  - St Thomas Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - St Mary's Hospital - Imperial College Healthcare NHS Trust, Hammersmith Hospital . Du Cane Road, London
  - The James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Schymik G, Lefevre T, Bartorelli AL, Rubino P, Treede H, Walther T, Baumgartner H, Windecker S, Wendler O, Urban P, Mandinov L, Thomas M, Vahanian A. European experience with the second-generation Edwards SAPIEN XT transcatheter heart valve in patients with severe aortic stenosis: 1-year outcomes from the SOURCE XT Registry. JACC Cardiovasc Interv. 2015 Apr 27;8(5):657-69. doi: 10.1016/j.jcin.2014.10.026. PMID 25946437